CLINICAL TRIAL: NCT02252562
Title: Reduction in 30-Day Postoperative Healthcare-Associated Infections Through Use of a Novel Hand Hygiene System
Brief Title: Hand Hygiene and Hospital Acquired Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Sage Products, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew Koff, Assistant Professor of Anesthesiology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D13081
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Complication of Surgical Procedure
Keywords: Hand hygiene; Hospital acquired infections (HAI); Healthcare acquired infections (HCAI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard practice (No Intervention): Usual intraoperative hand hygiene (standard wall mounted devices and machine and/or cart based dispensers)
- Personal hand hygiene device (Experimental): Intraoperative use of personalized body worn alcohol dispensers incorporating a novel wireless tracking system [(SAGE Products Inc., Cary, Il),
  Interventions: Device: Sage Personal Hand Hygiene System

INTERVENTIONS:
Device: Sage Personal Hand Hygiene System — Utilization of a health care provider worn personal hand hygiene system during routine practice in the intra-operative setting with provider specific individual feedback.
  Arms: Personal hand hygiene device

SUMMARY:
Healthcare-associated infections (HCAIs) and evolving bacterial resistance are major public health concerns that impact all areas of healthcare. Further work is needed to better understand these healthcare issues so that effective preventive measures can be developed.

The investigators have developed and validated an experimental model for studying the risk factors for bacterial cross contamination in the surgical operating room. The investigators have confirmed in our previous work that intraoperative bacterial transmission events occur frequently both within and between surgical cases and that these transmission events are linked to 30-day postoperative HCAIs and increased patient mortality.

In response, the investigators have implemented various strategies designed to bacterial transmission in the operating room, including anesthesia provider hand hygiene compliance. The investigators' recent work in the intensive care unit suggests that the hand hygiene system the investigators have previously studied could be further optimized.

The investigators now propose to evaluate the effectiveness of a multimodal hand hygiene system enhanced with novel wireless technology designed to facilitate real-time group and individual performance feedback.

The investigators hypothesize that the use of this system will increase hourly hand decontamination events of anesthesia and circulating nurse providers and reduce 30-day postoperative healthcare-associated infections HCAIs (primary outcome), reduce hospital stay duration, and hospital re-admission rates, and mortality(secondary outcomes).

DETAILED DESCRIPTION:
Healthcare-associated infections (HCAIs) and evolving bacterial resistance are major public health concerns that impact all healthcare arenas. Further work is indicated to better understand these healthcare issues in order that effective preventive measures can be developed.

The investigators have developed and validated an experimental model for studying the mechanisms, risk factors for, and implications of bacterial cross contamination in the surgical operating room. The investigators have confirmed through use of this model that intraoperative bacterial transmission events occur frequently within and between operative cases and that these transmission events are linked to 30-day postoperative HCAIs and to increased patient mortality. In response, the investigators have implemented and evaluated various strategies designed to target risk factors for intraoperative bacterial transmission events including anesthesia provider hand hygiene compliance, improved handling and design of intravascular catheters, and improved environmental decontamination of high-risk objects. While these focused strategies have been successful in reducing transmission events and the incidence of 30-day postoperative infections, the investigators' recent work in the intensive care unit suggests that the hand hygiene system the investigators studied could be further optimized. The investigators now propose to evaluate the effectiveness of a multimodal hand hygiene system enhanced with novel wireless technology designed to facilitate real-time group and individual performance feedback, two evidence-based educational interventions, in reducing 30-day postoperative HCAIs (primary outcome) and intraoperative bacterial transmission events, hospital stay duration, and hospital re-admission rates (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

1. Operating room environments involving adult patients undergoing general anesthesia, according to usual practice, for elective or urgent and emergent orthopedic, plastic, neurosurgical, cardiothoracic, urological, general abdominal, gynecological, vascular, or ear/nose/and throat surgical procedures
2. Requirement of a peripheral and/or central intravenous catheter

Surgical inclusion procedures were selected because they captured the majority of 30-day postoperative infections in a prior multi-center study that we conducted across three major academic medical centers [3].

The investigators will [randomize by the day in order to ensure that the treatment and control arms maintain their integrity and to facilitate an environment conducive to behavior change.] The investigators anticipate that the randomization strategy will allow equal distribution of urgent and emergent patients in the treatment and control groups. Patients with a prior infection and/or preexisting decolonization will be included and will be expected to be equally distributed between study groups given the randomized study design. For HCAI analysis, only new infection sites and/or a different organism of infection will be considered a new HCAI, per NHSN definitions (see below). The investigators realize that decolonization procedures have the capacity to reduce the effect size, and as such, we have appropriately adjusted the sample size (see statistical section).

Exclusion Criteria:

1. Pediatric patients
2. Lack of an intravenous catheter
3. Pregnant
4. A surgical procedure outside of the classes listed above
5. Adjustments on the day of surgery given the following considerations:

   * Provider allergy/intolerance to 64% alcohol: In the case where the primary anesthesia provider conveys a prior allergy to 64% alcohol and/or a history of significant contact dermatitis, the operating room will be excluded from enrollment. If a primary anesthesia provider develops an allergy and/or contact dermatitis during the study period, this will be documented, and operating rooms assigned to the primary anesthesia provider for future cases will be excluded. The expectation will be that all key providers working in operating rooms randomized to the intervention will participate in utilization of the device. If an operating room is randomized and a provider subsequently refuses to participate for any reason, the operating room will be excluded from the primary analysis but included in an intention-to-treat analysis. An additional operating room will be randomized for each such occurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3256 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen O Heard, MD, Study Chair — UMass Memorial Health
Locations (2):
- United States (2):
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Background] Koff MD, Loftus RW, Burchman CC, Schwartzman JD, Read ME, Henry ES, Beach ML. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a novel device. Anesthesiology. 2009 May;110(5):978-85. doi: 10.1097/ALN.0b013e3181a06ec3. PMID 19352154
- [Background] Loftus RW, Koff MD, Burchman CC, Schwartzman JD, Thorum V, Read ME, Wood TA, Beach ML. Transmission of pathogenic bacterial organisms in the anesthesia work area. Anesthesiology. 2008 Sep;109(3):399-407. doi: 10.1097/ALN.0b013e318182c855. PMID 18719437
- [Result] Koff MD, Brown JR, Marshall EJ, O'Malley AJ, Jensen JT, Heard SO, Longtine K, O'Neill M, Longtine J, Houston D, Robison C, Moulton E, Patel HM, Loftus RW. Frequency of Hand Decontamination of Intraoperative Providers and Reduction of Postoperative Healthcare-Associated Infections: A Randomized Clinical Trial of a Novel Hand Hygiene System. Infect Control Hosp Epidemiol. 2016 Aug;37(8):888-895. doi: 10.1017/ice.2016.106. Epub 2016 Jun 7. PMID 27267310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Operating room enrollment occurred from September 30, 2013, to June 17, 2014, at Dartmouth-Hitchcock Medical Center and from January 8, 2014, to August 21, 2014, at UMass Memorial Medical Center. Five to 10 operating rooms were enrolled Monday-Friday for each of 20 working days per month at each site.
Pre-assignment Details: The randomization unit was the operating room (OR); not the patient or provider. Clinicians were educated on the purpose of the study and utilized standard practice or hand hygiene device based on the ORs. 316 clinicians utilizing the personal hand hygiene device were followed for assessment, but not enrolled.
Units Other Than Participants: Operating Rooms
Period: Overall Study
Arm/Group | Standard Practice | Personal Hand Hygiene Device
Started (Operating rooms) | 1620; 1620 Operating Rooms | 1636; 1636 Operating Rooms
Completed (Operating rooms) | 1620; 1620 Operating Rooms | 1636; 1636 Operating Rooms
Not Completed | 0; 0 Operating Rooms | 0; 0 Operating Rooms

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are the patients who were seen in the operating rooms. Clinicians were not enrolled in the study and baseline data was not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Practice | Personal Hand Hygiene Device | Total
Number analyzed (Participants) | 1620 | 1636 | 3256
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.29 (16.4) | 56.75 (16.6) | 57.02 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 814 | 785 | 1599
  Male | 806 | 851 | 1657
Region of Enrollment [Number; unit: participants]
  United States | 1620 | 1636 | 3256

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Healthcare Acquired Infections
Description: Patients with a prior infection and/or preexisting decolonization will be included and will be expected to be equally distributed between study groups given the randomized study design. For HCAI analysis, only new infection sites and/or a different organism of infection will be considered a new HCAI, per NHSN definitions.
Time Frame: 30-day after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Practice | Personal Hand Hygiene Device
Number analyzed (Participants) | 1620 | 1636
Participants | 108 | 116
Statistical Analysis 1: Comparison: Standard Practice vs Personal Hand Hygiene Device; Test type: Equivalence — We hypothesized a potential 66% reduction from a baseline incidence of 0.16 on the basis of prior interventions, but we assumed for power considerations a more conservative reduction of 40% from a baseline incidence of 0.12 averaged across all patients in each arm. Assuming a 10% loss to follow-up, we required 1,600 patients per group for a power of 0.9 with a type 1 error of .05; fixed effects univariable analysis; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.82 to 1.40]

2. Secondary Outcome: Hospital Re-admission Rates
Description: Readmission to the hospital within 30 days of discharge
Time Frame: Within 30 days of discharge
Population: Data was not collected.
Arm/Group | Standard Practice | Personal Hand Hygiene Device
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mortality
Description: Patient Mortality
Time Frame: Within 30 Days of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Practice | Personal Hand Hygiene Device
Number analyzed (Participants) | 1620 | 1636
Participants | 6 | 7

4. Secondary Outcome: Hospital Duration
Description: Duration of Hospital Stay
Time Frame: 30 days after surgery
Population: Data was not collected
Arm/Group | Standard Practice | Personal Hand Hygiene Device
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Hand Hygiene Events Per Hour Utilizing the Device
Description: The number of times non-scrubbed personnel (anesthesia providers and circulating nurses) perform hand hygiene during OR cases for the treatment group.
Time Frame: During active OR cases
Population: A control arm was not tabulated as the control group did not utilize the study device.
Measure: Mean (Standard Deviation); unit: hand decontamination event per hour
Groups:
- Clinicians: Clinicians who were observed in for the Treatment arm utilizing the study device
Arm/Group | Clinicians
Number analyzed (Participants) | 316
hand decontamination event per hour | 4.3 (2.9)

ADVERSE EVENTS:
Time Frame: 30 days postoperative
Description: Adverse events related to the study outcome measures (Health-care-associated infections) were collected for patients only. AE's were not collected for clinicians.
Arm/Group | Standard Practice | Personal Hand Hygiene Device
All-Cause Mortality (participants affected / at risk) | 6/1620 | 7/1636
Serious Adverse Events (participants affected / at risk) | 0/1620 | 0/1636
Other Adverse Events (participants affected / at risk) | 0/1620 | 0/1636

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes